CLINICAL TRIAL: NCT06476626
Title: Maternal Reflective Functioning During the Transition to Motherhood as a Protective Factor in the Relationship Between Personal and Environmental Characteristics and the Mental Health of Both the Mother and the Infant
Brief Title: Maternal Reflective Functioning During the Transition to Motherhood
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Yael Enav, Head of Emotional Regulation and Mentalization Lab, University of Haifa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 086/24
Record Dates: First submitted 2024-06-06; First posted 2024-06-26 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Pregnancy; Primiparous Women
Keywords: pregnancy; primiparous women; anxiety; depression; stress; mentalization; reflective function
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maternal Reflective Functioning intervention group (Experimental): Will participate in a 4 session online psycho-educational workshop during pregnancy and after birth, focused on MRF.
  Interventions: Other: Maternal Reflective Function Workshop
- Wiat-list control group (No Intervention): group will undergo same measurements points with no intervention

INTERVENTIONS:
Other: Maternal Reflective Function Workshop — 4 session group online intervention focused on psycho-educational knowledge regarding emotional regulation and specifically MRF. group size- up to 15 participants. 2 sessions will be during pregnancy and 2 sessions will taken place 1 and 3 months after birth.
  Arms: Maternal Reflective Functioning intervention group

SUMMARY:
The goal of this clinical trial is to learn about Maternal Reflective Function (MRF) during the transition to motherhood. The main questions it aims to answer are:

Does MRF mediates the connection between risk factors for mental health difficulties during first pregnancy and motherhood (the transition to motherhood) and outcomes related to the mother, the infant, and their relationship.

Participants will:

Answer questionnaires and clinical interviews during pregnancy and after birth of the first child (twice at third trimester, 1 and 3 months after birth).

intervention group will participate in an online short intervention to enhance MRF.

DETAILED DESCRIPTION:
Using this trial, the investigators will be able to better understand rather MRF moderate the connection between risk factors to outcomes after birth related to both the mother and the infant. Using RCT design we will be able to understand mechanism of change.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women in 27-30 weeks pregnant in enrollment
* speak read and understand Hebrew
* Has a connection to internet and ZOOM platform.
* Ready to participate in a group workshop

Exclusion Criteria:

* Women who can't participate in a online workshop due to physical or mental health difficulties.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — the Workshop aimed to primiparous during the transition to motherhood.
Enrollment: 200 (Estimated)
Dates: Start 2024-07-15 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Maternal Reflective Functioning questionnaires | Twice in third trimester of pregnancy (Before and after intervention), 1 and 3 months after birth.
  Will be measured using Parental Reflective Function questionnaires for pregnancy P-PRFQ (Pajulo et al., 2015) and after birth (Parental Reflective Functioning Questionnaire PRFQ, Luyten et al., 2017). Likert Scale from 1 (Greatly disagree) to 7 (Greatly agree).
Maternal Reflective Functioning interviews | Once in third trimester of pregnancy ,1 months after birth.
  Will be measured using Pregnancy Interview (PI, Slade et al., 1987; Slade, 2003) before labor, and Parental Developmental Interview (PDI-R2 short form, Slade et al., 2003) after labor. Reflective Function Coding Scale- from -1 (No Reflective Function) to 9 (Very high Reflective Function)

SECONDARY OUTCOMES:
Depression. | Third trimester of pregnancy, 1 and 3 months after birth.
  depression level before, during and after pregnancy and birth, using Edinburgh Postnatal Depression Scale (EPDS, Cox, Holden, & Sagovsky, 1987). Likert Scale from 1 (Most of the time) to 4 (Almost never).
Anxiety | Third trimester of pregnancy, 1 and 3 months after birth.
  Anxiety level before, during and after pregnancy and birth using Depression Anxiety Stress Scale (DASS-21 short form, Lovibond & Lovibond, 1995 ). Likert Scale from 0- Does not describe my situation at all, to 3- Describes my situation very much.
Exposure to traumatic life events | At enrollment.
  exposure to ongoing war and political violence in the region using Political Life Events (PLE; Based on Slone et al., 1997, elaborated and adjusted by Yael Meir & Yael Enav, 2024, not published). Yes/No question and if Yes answered- Likert Scale from 1- Not at all to 5- Very much.
Social Support | Third trimester of pregnancy, 1 and 3 months after birth.
  Social support before and during pregnancy using Multidimensional Scale of Perceived Social Support (MSPSS, Zimet et al., 1988). Likert Scale from 1- Very agree, to 7- Very disagree.
Relationship satisfaction | Third trimester of pregnancy, 1 and 3 months after birth.
  Relationship satisfaction before and during pregnancy using Couple satisfaction index (CSI-16, Funk & Rogge, 2007). Likert Scale from 0- Not true at all, to 5- Very true.
High risk pregnancy | At enrollment.
  Medical high risk during pregnancy using a single question in initial demographic and personal details questionnaire.
Cognitive bias | Third trimester of pregnancy, 3 months after birth.
  Cognitive bias before, during and after pregnancy and birth using an go-no-go, infants expression interpretation, and focus of attention assignments.
Mother-infant bonding | Third trimester of pregnancy, 1 and 3 months after birth.
  Mother-infant bonding before birth using Prenatal Attachment Inventory (PAI: Muller & Mercer, 1993) after birth using Postpartum Bonding Questionnaire (PBQ, Brockington et al, 2006 ). PAI Likert Scale from 1- Almost never, to 4- Almost always.
Mother Emotional Regulation | Third trimester of pregnancy, 1 and 3 months after birth.
  Measured using Emotional Regulation Questionnaire (ERQ, Gross & John, 2003). Likert Scale from 1- Strongly disagree to 7- Strongly agree. PBQ Likert Scale from 1- Never to 6- Always
Infant weight | 1 and 3 months after birth.
  Gain of weight using a single question regarding infant's weight.
Maternal self-efficacy | 1 and 3 months after birth.
  Measured using Maternal self-efficacy Scale (Kestler-Peleg et al., 2015). Likert Scale from 1- Not at all, to 4- Very much.
Quality of sleep | 1 and 3 months after birth.
  Quality of sleep using Brief Infant Sleep Questionnaire (BISQ; Sade, 2004). Likert Scale from 1- Not at all to 4- Usually.

CONTACTS AND LOCATIONS:
Overall Officials: Yael Enav, Phd, Principal Investigator — University of Haifa
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
All IPD excluding personal information given by participants in interview (records and transcripts), however coded information for these interview will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available starting from 1 year after publishing of the primary results, with no limitation on duration of access.
Access Criteria: 1. Eligibility*: Access restricted to researchers affiliated with accredited academic institutions or healthcare organizations with relevant credentials.
  2. *Application*: Submit application form, research proposal, and CV to the principal investigator or designated contact.
  3. *Review and Approval*: Applications reviewed by the data access committee. Decision within 4-6 weeks.
  4. *Conditions of Use*: Data to be used solely for the approved project. Maintain confidentiality and data security. No third-party sharing without approval.
  5. *Publication and Reporting*: Submit summary of findings within 12 months. Acknowledge original study in publications and provide copies to the principal investigator.
URL: https://drive.google.com/drive/folders/1Z1JQq09fUMfCG6AHNM_4WLdIQLGYcTOW?usp=drive_link